CLINICAL TRIAL: NCT02715570
Title: A Randomised, Single-blind, Placebo-controlled, Study to Assess the Safety and Tolerability of Single Escalating and Repeat, Inhaled Doses of PC945 in Healthy Subjects Combined With a Randomised, Single-blind, Placebo-controlled, Parallel Group to Assess the Safety and Tolerability of a Single Dose of Inhaled PC945 in Subjects With Mild Asthma
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of PC945
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PC_ASP_001; 2015-003327-64 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Aspergillosis
Keywords: Aspergillus species; Filamentous fungi; 14-alpha Demethylase Inhibitors; Anti-Infective Agents; Antifungal Agents; Enzyme Inhibitors; Aspergillosis; Allergic Bronchopulmonary; Asthma
MeSH Terms: conditions — Aspergillosis; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose - healthy volunteers (Experimental)
  Interventions: Drug: PC945 - single doses; Drug: Placebo - single doses
- Repeat dose - healthy volunteers (Experimental)
  Interventions: Drug: PC945 - repeat doses; Drug: Placebo - repeat doses
- Single dose - asthmatic patients (Experimental)
  Interventions: Drug: PC945 - single doses; Drug: Placebo - single doses

INTERVENTIONS:
Drug: PC945 - single doses — Safety and tolerability of single doses
  Arms: Single dose - asthmatic patients; Single dose - healthy volunteers
Drug: Placebo - single doses — Safety and tolerability of single doses
  Arms: Single dose - asthmatic patients; Single dose - healthy volunteers
Drug: PC945 - repeat doses — Safety and tolerability of repeat doses
  Arms: Repeat dose - healthy volunteers
Drug: Placebo - repeat doses — Safety and tolerability of repeat doses
  Arms: Repeat dose - healthy volunteers

SUMMARY:
PC945 is a new medicine being developed for treatment of fungal lung diseases. The main purpose of this study is to investigate the safety, tolerability and pharmacokinetics of single and repeat doses of PC945

ELIGIBILITY:
Inclusion Criteria:

All subjects (Cohorts 1, 2 & 3)

* Male or female, aged between 18 and 65 years inclusive (at the time of consent) who fit one of the following criteria: Women of childbearing potential who are willing and able to use required contraception from screening until 30 days after receipt of the final dose; Women of non-childbearing potential defined as being amenorrhoeic or have been permanently sterilised; Men who are willing and able to use required contraception from the time of the first dose, until 90 days after receipt of the final dose of study medication.
* Females with a negative pregnancy test at screening and at Day -1.
* Willing and able to adhere to the restrictions and prohibitions required by this protocol.
* Signed informed consent form.
* Body weight ≥ 50 kg and body mass index (BMI) within the range 18 - 30 kg/m2 (inclusive).
* Average QTcF <450 msec at screening and pre-dose.
* Vital signs assessments within normal ranges

Healthy Subjects (Cohorts 1 and 2)

* Healthy as determined by a physician based on a full medical examination.
* Spirometry readings (FEV1 and FVC) to be ≥ 80% of predicted value and FEV1/FVC ratio > 0.7 at screening.

Subjects with Asthma (Cohort 3)

* Diagnosis of asthma.
* Positive result to methacholine challenge at the screening visit.
* FEV1 >60% of predicted normal value at screening.
* Stable asthma based on physician assessment at screening, with no changes of therapy in the 12 weeks prior to screening and no hospitalization or visit to accident and emergency for asthma in the 12 months prior to screening
* Otherwise healthy on the basis of a full medical examination at screening

Exclusion Criteria:

All subjects (Cohorts 1, 2 & 3)

* Any acute illness.
* Upper or lower respiratory tract infection within 4 weeks of the screening visit or randomisation.
* Use of prescription medications within 14 days of the Screening visit.
* Taking over the counter (OTC) medications other than vitamins or multivitamins, within 14 days prior to Screening.
* History of regular alcohol consumption within 6 months of the study with average weekly intake of >21 units for males, or >14 units for females.
* History of drug or alcohol abuse within the previous 5 years.
* Smoker (regular or irregular), or has smoked or used nicotine-containing products (including e-cigarettes) within the 6 months prior to screening or has a smoking history of ≥ 10 pack years.
* Positive test for HIV-1 & -2 antibodies at screening.
* Positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result at screening.
* Positive test for alcohol, smoking or drugs of abuse at screening or Day -1.
* Received an experimental drug or used an experimental medical device within last 3 months.
* Allergy to any of the active or inactive ingredients in the study medication.
* Donation of blood in excess of 500 mL within a 3 month period prior to dosing, or if study participation would result in blood loss in excess of 500 mL in a 3 month period.
* Mentally or legally incapacitated.
* An employee of the Sponsor or contract research organisation (CRO), or a relative of an employee of the Sponsor or CRO.
* Unable or unwilling to undergo multiple venepuncture procedures or poor access to veins suitable for cannulation.
* Pregnant or lactating female

Healthy subjects (Cohorts 1 and 2)

* Any chronic illness or clinically relevant abnormality identified on the screening medical assessment, laboratory tests or ECG.

Subjects with asthma (Cohort 3)

* Had an episode of life-threatening asthma.
* Presence of clinically significant diseases other than asthma, hyper-responsive airways, seasonal allergic rhinitis or atopic diseases.
* Experienced an acute asthma exacerbation in the 12 months prior to screening requiring hospitalisation or accident and emergency treatment or management with systemic or injectable steroids.
* Uncontrolled, or moderate to severe asthma based on PI assessment and/or use of prohibited medications, or has required treatment with these therapies in the previous 12 weeks.
* History or presence of any known conditions contraindicated for methacholine challenge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Cohort 1 - 12 weeks; Cohort 2 - 7 weeks; Cohort 3 - 6 weeks
  Assessment of number of adverse events reported by subjects following dosing
12-lead ECG assessment | Cohort 1 - 12 weeks; Cohort 2 - 7 weeks; Cohort 3 - 6 weeks
  Change from pre-dose values
Vital signs assessment (blood pressure and heart rate - measured together) | Cohort 1 - 12 weeks; Cohort 2 - 7 weeks; Cohort 3 - 6 weeks
  Change for pre-dose values
Clinical laboratory assessments (blood and urine samples - measured together) | Cohort 1 - 12 weeks; Cohort 2 - 7 weeks; Cohort 3 - 6 weeks
  Change from pre-dose values
Spirometry assessment (FEV1 & FVC - measured together) | Cohort 1 - 12 weeks; Cohort 2 - 7 weeks; Cohort 3 - 6 weeks
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma concentration data of PC945 | Cohort 1 (4 treatment periods) & Cohort 3 (1 treatment period) Day1 = 8 samples; Day2 = 2 samples; Day3 = 1 sample; F/U = 1 sample. Cohort 2 - Days1&7 = 10 samples; Days2,5,6 = 1 sample; Day8 = 2 samples; Day9 = 1 sample; F/U = 1 sample
  Blood levels of PC945 measured after dosing
Spirometry assessment (FEV1) | Cohort 3 only - Day 1, 8 hours
  Observed drops in FEV1 assessment after dosing patients with mild asthma

OTHER OUTCOMES:
Determination of exogenous fungal flora | Cohort 1 (4 treatment periods) & Cohort 3 (1 treatment period) Day1 = 1 sample; Day3 = 1 sample. Cohort 2, Day 1 = 1 sample; Day 9 = 1 sample
  Assessment of fungal flora found in mouth and throat after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, FFPM, MSc, Principal Investigator — cro
Locations (1):
- Parexel EPCU, Harrow, Middlesex, United Kingdom